CLINICAL TRIAL: NCT01842919
Title: Dance and Huntington Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C12-64; 2012-A01669-34 (Registry Identifier: IRDB)
Record Dates: First submitted 2013-04-03; First posted 2013-04-30 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2017-09

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Huntington patient (Other): This group will perform Magnetic Resonance Imaging (MRI), kinesthetic test and psychological questionnaires before and after 8 months of dance lessons
  Interventions: Other: Kinesthetics tests; Other: Psychological questionnaires; Other: structural Magnetic ResonanceImaging (MRI)
- Assisting Person (Other): This group will perform MRI, kinesthetic test and psychological questionnaires before and after 8 months of dance lessons
  Interventions: Other: Kinesthetics tests; Other: Psychological questionnaires; Other: structural Magnetic ResonanceImaging (MRI)
- Pilot subject (Other): Healthy volunteers to set up the kinesthetic test
  Interventions: Other: Kinesthetics tests

INTERVENTIONS:
Other: Kinesthetics tests
Other: Psychological questionnaires
  Arms: Assisting Person; Huntington patient
Other: structural Magnetic ResonanceImaging (MRI)
  Arms: Assisting Person; Huntington patient

SUMMARY:
In this project investigators will evaluate the benefits of contemporary dance training using a comprehensive test battery combining standard neuropsychological batteries, psychological questionnaires on emotion, empathy and quality of life, structural magnet-resonance tomography (MRI), as well as psychophysical tests on movement recognition and agency, the sense of being in control of one's own movement.

For 10 years now two experienced dancer-choreographers lead dance workshops for people with Huntington's Disease (HD) and their family and caregivers in Paris. This project will evaluate objectively the effects these workshops have, by assessing a new group of 18 patients and their partners and caregivers before and after 8 month of weekly dance training.

People with HD are troubled by involuntary movements, of which they are however not accurately aware, but moreover they become impaired at recognising instrumental actions in others. It is well known that observing somebody else's action and executing the same action rest on a common neural network. This might mean that improving one's own action execution can improve the observation and understanding of others' actions in turn. Here, investigators will investigate both the impact the movement impairments caused by HD might have on patients themselves as well as on their partners and caregivers, as a consequence of the fact that own and other action representations are shared. After 8 months of contemporary dance training, both groups will be tested again, in order to establish if both action execution (self) and perception (in others) have improved.

Other recent psychophysics and brain imaging experiments have demonstrated how the sense of agency is composed from external cues (for example sound) of the consequences of movements, and from internal sensorimotor information that result from the action plan. Importantly, in HD the latter input might be impaired, but this has never been systematically tested. Making use of a psychophysics paradigm disentangling the two cues to agency investigators first monitor the sense of their own movement in HD, and further assess the changes in agency and in the role of these cues to agency after eight months of contemporary dance practice.

Finally investigators will monitor the structural brain changes accompanying this progress, comparing the brain before and after regular dance practice and correlating action recognition psychophysics measures of agency with these changes.

In sum, this project has a double impact. Firstly it will scientifically evaluate the impact of dance on the normal but especially the brain affected by a neurodegenerative disease that causes movement impairments, and establish its effect on behaviour and wellbeing. Secondly it will evaluate in patient partners and caregivers how they represent the patients' as well as their own movements and how this changes with dance practice.

ELIGIBILITY:
Inclusion Criteria:

Huntington patient

* Patients with Huntington's disease (documented by a genetic test.)
* Ability and intention to follow the dance workshop of the association Micadanse once a week for 8 months (Total Functional Capacity score (TFC) > 10).
* Have an assisting person who also lends him/herself to the protocol.
* Showing no indications against to the achievement of MRI.

Assisting person:

* No history of neurological or psychiatric disorders.
* Showing no indications against to the achievement of MRI.

Exclusion Criteria:

* Have already taken dance lessons.
* Neurological or psychiatric history.
* Inability to achieve MRI
* History of significant head injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-07-28 (Actual); Study Completion 2016-07-08 (Actual)

PRIMARY OUTCOMES:
Detection score | Day 1
  The subject performs movements imposed which are recorded by sensors in the form of bright spots.
  It shows the participant of "bright spots" of himself or of another subject of the same sex and must indicate whether of himself or another person.
  The number of correct answers is calculated and subtracted from the numbers of false positives.
Detection score | 9th month
  The subject performs movements imposed which are recorded by sensors in the form of bright spots.
  It shows the participant of "bright spots" of himself or of another subject of the same sex and must indicate whether of himself or another person.
  The number of correct answers is calculated and subtracted from the numbers of false positives.
  The number of correct answers is calculated and subtracted from the numbers of false positives.

REFERENCES:
- [Result] Trinkler I, Chehere P, Salgues J, Monin ML, Tezenas du Montcel S, Khani S, Gargiulo M, Durr A. Contemporary Dance Practice Improves Motor Function and Body Representation in Huntington's Disease: A Pilot Study. J Huntingtons Dis. 2019;8(1):97-110. doi: 10.3233/JHD-180315. PMID 30776016